CLINICAL TRIAL: NCT01858259
Title: Prevention and Treatment of Interstitial Lung Disease in Systemic Sclerosis
Brief Title: Treatment and Prevention of Progression of Interstitial Lung Disease in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gabriela Riemekasten (Other)
Collaborators: European Union (Other); University of Giessen (Other); University of Zurich (Other); University of Paris 5 - Rene Descartes (Other); University of Florence (Other); University of Campania Luigi Vanvitelli (Other); University of Basel (Other); University College, London (Other); Charite University, Berlin, Germany (Other); University of Pecs (Other); University of Leeds (Other); Schoen Klinik Hamburg Eilbek (Other)
Responsible Party: Sponsor-Investigator, Gabriela Riemekasten, Prof. Dr. med. Gabriela Riemekasten, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: HEALTH-F5-2012-305495-OT3
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Systemic Sclerosis; Interstitial Lung Diseases
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- cyclophosphamide: Patients receiving cyclophosphamide
- azathioprine: Patients receiving azathioprine
- mycophenolate mofetil: Patients receiving mycophenolate mofetil
- methotrexate: Patients receiving methotrexate
- no therapy: Patients receiving no immunosuppressive therapy

SUMMARY:
Systemic sclerosis (SSc) is an orphan, multiorgan disease affecting the connective tissue of the skin and all internal organs. Interstitial lung disease is a frequent morbidity and mortality-driving manifestation in systemic sclerosis.

This observational trial (OT) is part of the collaborative project "DeSScipher", one out of five OTs to decipher the optimal management of systemic sclerosis. Aim of this observational try is to identify:

* The state of clinical practice in Europe for prevention and treatment of interstitial lung disease and its impact on lung function and disease progression
* The potential predictors and confounders for response to therapy

DETAILED DESCRIPTION:
Patients are routinely evaluated every 3 months over a 12-months period by medical history, physical examination, pulmonary function tests, VAS lung score and SF-36, SHAQ. Also, their medication and possible medication changes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis fo SSc according to the ACR/EULAR criteria for adult or the PRES/ACR/EULAR criteria for juvenile SSc patients
* SSc patients with proven ILD (by X-ray or CT scan)
* Treatment with standard dosages according to current practice with (i) cyclophosphamide, (ii) azathioprine, (iii) mycophenolate mofetil, (iv) methotrexate, or (v) no therapy

Exclusion Criterion:

* Patients with previous exposure to silica or asbestos

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are adult and juvenile SSc patients from the EUSTAR cohort (MEDSonline database) and the jSScWG cohort
Sampling Method: Probability Sample
Enrollment: 1372 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with 10% decline in FVC | 1 year
  The proportion of patients with ILD progression as defined by a 10% decline in FVC within 1 year of therapy

SECONDARY OUTCOMES:
The time to a 15% decline in DLCO or a drop <55% of predicted lung function | 1 year
The mortality due to lung fibrosis | 1 year
The need for oxygen support | 1 year

OTHER OUTCOMES:
Identification of confounders | 1 year
  Parameters with impact on ILD progression independent of therapies, such as SSc subgroups, presence of antibodies, presence of vasculopathy, time to therapy initiation, degree of lung fibrosis defined by FVC values, age at disease onset and at treatment initiation, gender, co-morbidities and other confounders.
Evaluation of the incidence of drug-related adverse events | 1 year
Evaluation of the incidence of withdrawal from treatment due to drug-related adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Riemekasten, Prof., Principal Investigator — Charité Universitätsmedizin Berlin, Charité Centrum 12 für Innere Medizin und Dermatologie, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie; Christopher Denton, Prof., Principal Investigator — Royal Free Hospital, University College London London; Ulf Müller-Ladner, Prof., Study Chair — Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology
Locations (11):
- Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM 1016, Paris, France
- Germany (3):
  - Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Charité Centrum 12 für Innere Medizin und Dermatologie, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Centre for Pediatric Rheumatology, Klinikum Eilbek, Hamburg
- Pecsi Tudomanyegyetem - University of Pecs, Pécs, Hungary
- Italy (2):
  - University of Florence, Denothe Centre, Division of Rheumatology AOUC, Department of Biomedicine, Florence
  - Policlinico, Via Pansini, Napoli-Italia
- Switzerland (2):
  - Felix-Platter Spital, University of Basel, Basel
  - University of Zurich, Department of Rheumatology, Zurich
- United Kingdom (2):
  - The Universitiy of Leeds, Division of Rheumatic and Musculoskeletal Disease, St James's University Hospital, Leeds
  - Royal Free Hospital, University College London, London